CLINICAL TRIAL: NCT06685575
Title: Comparative Outcomes of Conventional Transforaminal Lumbar Interbody Fusion With Posterior Decompression Surgery Versus Endoscopic Foraminotomy Surgery in Stable Lumbar Foraminal Stenosis An Ambi-directional Cohort Study
Brief Title: Comparative Outcomes of Conventional TLIF With Posterior Decompression Surgery Versus Endoscopic Foraminotomy Surgery
Acronym: TLIF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 020/2567
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Foraminal Stenosis
Keywords: Lumbar Foraminal Stenosis; endoscopic decompression surgery; Endoscopic Foraminotomy Surgery; TLIF in lumbar foraminal stenosis; stable lumbar foraminal stenosis

STUDY DESIGN:
Intervention Model Description: Comparative Outcomes of Conventional Transforaminal Lumbar Interbody Fusion With Posterior Decompression Surgery Versus Endoscopic Foraminotomy Surgery in Stable Lumbar Foraminal Stenosis An Ambi-directional Cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Transforaminal Lumbar Interbody Fusion With Posterior Decompression Surgery (No Intervention): standard surgery for foraminal stenosis
- Endoscopic Foraminotomy Surgery (Experimental): The new type of surgery to treat lumbar foraminal stenosis which does not lead to instability of the spine
  Interventions: Procedure: Endoscopic Foraminotomy Surgery

INTERVENTIONS:
Procedure: Endoscopic Foraminotomy Surgery — Endoscopic Foraminotomy Surgery in Stable Lumbar Foraminal Stenosis
  Arms: Endoscopic Foraminotomy Surgery

SUMMARY:
Comparative Outcomes of Conventional Transforaminal Lumbar Interbody Fusion With Posterior Decompression Surgery Versus Endoscopic Foraminotomy Surgery in Stable Lumbar Foraminal Stenosis An Ambi-directional Cohort Study

DETAILED DESCRIPTION:
Backgrounds :

Lumbar foraminal stenosis is a condition in which a spinal nerve is entrapped in a narrow lumbar foramen in degenerative lumbar spinal disorders. The gold standard treatment of this condition has not been proposed yet. Several different techniques for this problem has been described, including foraminotomy, facetectomy, partial pediculectomy, fusion, and distraction instrumentation.Nowadays, due to the great advancement of the technology in endoscopy expanded the indication of endoscopic decompression from the central canal to the extraforaminal zone, Which was difficult to gain access from the mere microscope.

Objectives :

To compare outcomes between posterior decompression With conventional transforaminal lumbar interbody fusion (TLIF) and full-endoscopic foraminoplasty (FELF) in stable lumbar foraminal Stenosis

Methods :

This is an ambi-directional cohort study, In retrospective part conducted from JAN2019-JAN2024 in Queen Savang Vadhana Memorial Hospital and the prospective part conducted from AUG2024 - JUNE 2025, Thailand. 60 patients presented with stable lumbar foraminal stenosis were divided into posterior decompression with conventional transforaminal lumbar interbody fusion (TLIF) group ( N=30) and full-endoscopic lumbar foraminoplasty (FELF) group (N=30). Demographic data and pre-perioperative parameters were analyzed. For TLIF group , Standard procedure had been performed.

Posterior decompression, pedicle screws and interbody cage ( Mont blanc, Spineway, France) insertion under image intensifier ( BV Pulsera,Philips).For endoscopic foraminoplasty , uniportal stenoscope ( Vertebris ,Riwospine ) was used to perform endoscopic decompressive surgery. Post-operative outcome , for instance , Visual Analog Scale (VAS) and the Oswestry Disability Index (ODI) were recorded at preoperative, post-op day1, 3 month, 6 month and 1 year respectively. Other parameters such as estimated blood loss (EBL), length of hospital stay and post- operative complications were also recorded

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80
* Persist radiculopathy and sciatica pain
* Patient that was diagnosed Stable lumbar foraminal stenosis
* Failed conservative for at least 6 months
* Patients who willing to join the study

Exclusion Criteria:

* Patients with unstable lumbar foraminal stenosis
* Patient with spine infection or tumor or fracture
* Patient with BMD less than -2.5 or osteopenia
* Patient with inflammatory joint diseases who on steroids
* Patient who has undergo with surgery that inserted metals in back
* Unable to answer questionnaires
* Cannot tolerate surgery due to severe medical comorbidities

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability index (ODI) score post-operation at 12months | 12 months
  Oswestry disability index (ODI) questionnaire at 12 months postoperative. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound. Minimal clinical difference has been evaluated across numerous types of spinal surgery, and has been shown to vary significantly.

SECONDARY OUTCOMES:
Oswestry disability index (ODI) score post-operation at 6week, 3 months and 6 months | 6week, 3 months and 6 months
  Oswestry disability index (ODI) questionnaire at 6week, 3 months and 6 months. The final score/index ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound. Minimal clinical difference has been evaluated across numerous types of spinal surgery, and has been shown to vary significantly
visual analog scale (VAS) of pain both leg and back | 1day, 2 weeks, 6weeks, 3 months, 6 months and 12 months
  visual analog scale (VAS) of pain.A Visual Analogue Scale (VAS) score is interpreted by measuring the distance from the "no pain" end of a 100-mm line to a mark made by the patient to indicate their pain level. A higher score indicates greater pain intensity.
estimated blood loss (EBL) | perioperation
  intraoperative estimated blood loss (EBL) measure in milliliter. estimated blood loss is a reliable predictor of actual blood loss during orthopedic procedures.
operative time | perioperation
  operative time measure in minutes, usually 60-90 minutes
length of hospital stay | from 3 days to 1 week
  length of hospital stay
time return to work | through the study completion, an average of 1 year
  time return to work
postoperative complications | through the study completion, an average of 1 year
  postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Tanyasinee Soonthornthum, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No
Data was save inform of microsoft excel spreadsheet and SPSS file